CLINICAL TRIAL: NCT05765032
Title: An Open Label, Multicenter, Phase Ib/II Study of SHR-A1921 in Combination With Other Anti-cancer Agents in Patients With Advanced Solid Tumors
Brief Title: Study of SHR-A1921 in Combination With Other Anti-cancer Agents in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1921-201
Record Dates: First submitted 2023-02-14; First posted 2023-03-13 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1921 (Experimental): A1：SHR-A1921+Adebrelimab A2：SHR-A1921+Carboplatin A3：SHR-A1921+Cisplatin A4：SHR-A1921+Bevacizumab A5：SHR-A1921+Adebrelimab+Carboplatin A6：SHR-A1921+Adebrelimab+Cisplatin B1：SHR-A1921+Adebrelimab B2：SHR-A1921+Adebrelimab+Carboplatin/Cisplatin
  Interventions: Drug: SHR-A1921；

INTERVENTIONS:
Drug: SHR-A1921； — Drug: SHR-A1921 administered as an IV infusion Drug: Adebrelimab administered as an IV infusion Drug: Carboplatin administered as an IV infusion Drug: Cisplatin administered as an IV infusion Drug: Bevacizumab administered as an IV infusion

SUMMARY:
This research study is a multicentre phase Ⅰb/Ⅱ Study to evaluate the efficacy and safety of SHR-A1921 in combination with other anti-cancer agents in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-75 years;
2. Be able to provide fresh or archived tumour tissue.
3. Ph 1b: clinically or pathologically diagnosed advanced solid tumour . Ph II: Histologically or cytologically confirmed, advanced or metastatic non-small cell lung cancer
4. With at least one measurable lesion (in accordance with RECIST v1.1)
5. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
6. With a life expectancy ≥ 12 weeks.
7. Sufficient organ functions.
8. Women of childbearing potential (WOCBP) and Male subjects whose partner are women of childbearing potential must agree to use a reliable and valid contraceptive method.

Exclusion Criteria:

1. Untreated brain metastasis or accompanied by meningeal metastases, spinal cord compression.
2. Uncontrolled pleural effusion, pericardial effusion, or abdominal effusion with clinical symptoms.
3. Previous or co-existing malignancies other than cured basal cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of the breast (DCIS), papillary thyroid carcinoma, and other malignancies that have been adequately treated and cured for ≥3 years
4. Hypertension that can not be well controlled through antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg); previous hypertensive crisis or hypertensive encephalopathy.
5. with any active or known autoimmune disease
6. with active pulmonary tuberculosis infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Experienced Any Dose-Limiting Toxicity (DLT) over the DLT period. （Phase 1b） | up to 21 days of cycle 1
Determination of Recommended Phase II dose (RP2D) （Phase 1b） | Up to 21 days of cycle 1
Objective Response Rate as Assessed by the Investigator according to RECIST v1.1（Phase II） | From baseline to progressive disease or death (approximately 1 year)

SECONDARY OUTCOMES:
Objective Response Rate as Assessed by the Investigator according to RECIST v1.1e (Ph1b only), | From baseline to progressive disease or death (approximately 1 year)]
Duration of Response as Assessed by the Investigator according to RECIST v1.1 | From baseline to progressive disease or death (approximately 1 year)
Disease Control Rate as Assessed by the Investigator according to RECIST v1.1 | From baseline to progressive disease or death (approximately 1 year)
Time to Response as Assessed by the Investigator according to RECIST v1.1 | From baseline to progressive disease or death (approximately 1 year)
Progression-free Survival as Assessed by the Investigator according to RECIST v1.1 | From baseline to progressive disease or death (approximately 1 year)
Overall survival | approximately 12months after last patient enrolled.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute& Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided